CLINICAL TRIAL: NCT06519929
Title: A Pilot Study Comparing Three Analgesia Approaches for Rib Fractures
Brief Title: Analgesic Techniques for Rib Fractures
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRISID-2022-1186
Record Dates: First submitted 2024-07-16; First posted 2024-07-25 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Rib Fractures
MeSH Terms: conditions — Rib Fractures

STUDY DESIGN:
Intervention Model Description: 3-arm, parallel-group, randomized controlled trial
Who Masked: Outcomes Assessor
Masking Description: Participants, care providers, and investigators will not be blinded but outcome assessors will be unaware of group assignment when doing baseline assessments and when performing some post-randomization assessments, such as those at 30 and 90 days by phone call.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- ESP block with catheter using ropivacaine (bolus followed by continuous infusion) (Experimental)
  Interventions: Procedure: ESP block with catheter using ropivacaine (bolus followed by continuous infusion)
- Lidocaine bolus (1 mg/kg) and infusion starting at 1 mg/kg/h (Active Comparator)
  Interventions: Drug: Lidocaine bolus (1 mg/kg) and infusion starting at 1 mg/kg/h
- Standard care with multimodal analgesia and opioids (No Intervention)

INTERVENTIONS:
Procedure: ESP block with catheter using ropivacaine (bolus followed by continuous infusion) — A total of ropivacaine 75mg will be injected into the plane via the needle, followed by placement of a catheter 3-5 cm into the plane. A continuous infusion of ropivacaine 0.2% will be started at 8 mL/h and may be titrated up to a maximum of 10mL/h. Bolus doses of 5 mL using ropivacaine 0.2% will be permitted for breakthrough pain (pain score ≥ 7/10) and may be administered no more frequently than every 6 hours. Patients will be assessed for LAST twice daily by asking about tinnitus, perioral numbness, or metallic taste. Any patient who responds positively to these symptoms will have infusion stopped for 2 h and then restarted at a rate 2 mL/h lower. If the symptoms occur again, the catheter infusion will be stopped and the catheter removed. After the 72-hour study period the ESP catheter may remain in place if the patient has ongoing analgesia needs or if analgesia is controlled with oral medication the catheter may be removed at request of the treating team.
  Arms: ESP block with catheter using ropivacaine (bolus followed by continuous infusion)
Drug: Lidocaine bolus (1 mg/kg) and infusion starting at 1 mg/kg/h — A bolus of 1 mg/kg based on ideal body weight will be given over 10 minutes with a physician present and infusions will be started at 1 mg/kg/h based on IBW. Infusions will run continuously for the first 72 h and can be continued beyond that at the discretion of the treating team if pain persists. Patients will be assessed for LAST twice daily. Any patient with suspected LAST will have lidocaine infusion stopped and a lidocaine plasma level will be sent. If symptoms resolve, the lidocaine infusion can be restarted at a rate 25% lower. If pain is refractory to the lidocaine infusion and multimodal adjuncts, the infusion may be increased to a maximum of 1.5 mg/kg/h (during first 24 h only). The actual duration of the infusion as well as total lidocaine dose given in mg will be recorded. Stopping criteria for lidocaine will include the occurrence of new EKG changes for which an alternative explanation is not more likely as well as LAST symptoms.
  Arms: Lidocaine bolus (1 mg/kg) and infusion starting at 1 mg/kg/h

SUMMARY:
This study will be a 3-arm, parallel-group, randomized controlled trial comparing three analgesic techniques for rib fractures with a sample size of 24 patients (8 per group). Patients will be randomly assigned to one of the following three groups: 1) ESP block with catheter using ropivacaine (bolus followed by continuous infusion); 2) lidocaine bolus (1 mg/kg) and infusion starting at 1 mg/kg/h; or 3) standard care with multimodal analgesia and opioids.

Our specific aims are:

1. To compare the opioid use and pain ratings over the first 72 hours after enrollment.
2. To quantify the changes in vital capacity, oxygen requirement, and freedom from mechanical ventilation that result from the intervention.
3. To explore the impact of ESP blocks and lidocaine infusions on the development of chronic pain and post-discharge opioid use (exploratory).

Inclusion Criteria:

• Adult patients ≥ 55 years old who have sustained 3 or more unilateral rib fractures and are admitted to the hospital.

Exclusion Criteria:

* Allergy to amide local anesthetics, lidocaine, or ropivacaine
* Pregnancy
* Bilateral rib fractures
* Coagulopathy (INR > 1.5; PTT > 1.5 times ULN, or platelets < 75,000)
* Conduction block on EKG
* Total body weight < 40 kg
* Painful distracting injuries: acute thoracic spine fracture, severe traumatic brain injury or spinal cord injury, unstable pelvic fracture, open abdomen
* Spine fracture at the level of intended ESP block
* Infection near the ESP insertion site or active bacteremia or sepsis
* Any patient deemed a poor candidate for ESP block and/or lidocaine infusion will also be excluded

ELIGIBILITY:
Inclusion Criteria:

* ≥ 55 years old
* Sustained 3 or more unilateral rib fractures and are admitted to the hospital

Exclusion Criteria:

* Allergy to amide local anesthetics or any study medications
* Pregnancy
* Bilateral rib fractures
* Coagulopathy (INR > 1.5; platelets < 100,000)
* Conduction block on EKG
* Spine fracture at the level of intended ESP block
* Infection near the ESP insertion site or active bacteremia or sepsis
* Any patient deemed a poor candidate for ESP block and/or lidocaine infusion will also be excluded

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-09-23 (Actual); Primary Completion 2025-08-31 (Actual); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Opioid Use in oral morphine equivalents (OME) | 72 Hours
  This will include both IV and oral opioids. Opioids given via PCA will also be prospectively recorded and included.
Brief Pain Inventory - current pain subscale (0-10) | 0-72 Hours
  The Brief Pain Inventory (short form) - average of all "current pain" ratings).

SECONDARY OUTCOMES:
Daily opioid use | 30 Days
  The total daily opioid use will be recorded and converted to OMEs. The PDMP will be used to confirm if needed.
Daily opioid Use | 90 Days
  The total daily opioid use will be recorded and converted to OMEs. The PDMP will be used to confirm if needed.
Brief Pain Inventory | Days 1-3
  Average pain (0-10) - this is the average of the "average pain" scores
Brief Pain Inventory | Day 30
  Average pain (0-10)
Brief Pain Inventory | Day 90
  Average pain (0-10)
Vital capacity (mL) | Baseline prior to intervention
  Volume of air expired after a maximal inspiration in mL measured with spirometer
Vital capacity (mL) | Day 1
  Volume of air expired after a maximal inspiration in mL measured with spirometer
Vital capacity (mL) | Day 2
  Volume of air expired after a maximal inspiration in mL measured with spirometer
Vital capacity (mL) | Day 3
  Volume of air expired after a maximal inspiration in mL measured with spirometer
Duke Activity Status Index | Baseline prior to intervention
  Functional status assessment (0-60 with 60 representing the best function)
Short-form 12 | Baseline prior to intervention
  Functional status assessment (0-100 with 100 representing best function)
Short-form 12 | Day 30
  Functional status assessment (0-100 with 100 representing best function)
Short-form 12 | Day 90
  Functional status assessment (0-100 with 100 representing best function)
3D-CAM/CAM-ICU | Day 1
  Delirium assessment (yes or no)
3D-CAM/CAM-ICU | Day 2
  Delirium assessment (yes or no)
3D-CAM/CAM-ICU | Day 3
  Delirium assessment (yes or no)
Respiratory depression | Days 1-3
  Naloxone use
Epidural eligibility | Day 1
  Clinical judgment of physician
RibScore | Day 1
  Score includes: >= 6 ribs fractured, flail chest, bilateral fractures, first rib fracture, >= 3 displaced fractures, fracture in each anatomical area
Presence of perioral numbness | Day 1
  Patient self report
Presence of perioral numbness | Day 2
  Patient self report
Presence of perioral numbness | Day 3
  Patient self report
Presence of tinnitus | Day 1
  Patient self report
Presence of tinnitus | Day 2
  Patient self report
Presence of tinnitus | Day 3
  Patient self report
Presence of metallic taste | Day 1
  Patient self report
Presence of metallic taste | Day 2
  Patient self report
Presence of metallic taste | Day 3
  Patient self report

CONTACTS AND LOCATIONS:
Overall Officials: Eric Schwenk, MD, Principal Investigator — Thomas Jefferson University
Locations (1):
- Thomas Jefferson University Hospital, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No